CLINICAL TRIAL: NCT03034109
Title: Transcranial Direct Current Stimulation (tDCS) in Post-Stroke Working Memory Deficits
Acronym: TDCS-PSMWD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Negative interim analysis.
Sponsor: Stony Brook University (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Andrew Goldfine, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 986244
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Stroke; Cognitive Deficit; Cognitive Impairment; Short-Term Memory Impairment
Keywords: Transcranial Direct Current Stimulation; Stroke; Electric Stimulation Therapy; Prefrontal Cortex; Electroencephalography; Cognition; Neurological Rehabilitation; Memory; Working Memory; Attention; Concentration; Short-Term Memory; Planning; Executive Function; Cerebrovascular disease
MeSH Terms: conditions — Stroke; Cognition Disorders; Cognitive Dysfunction; Cerebrovascular Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- tDCS conventional stimulation (Experimental): Transcranial Direct Current Stimulation:
  The anode will be placed over the left dorsal lateral prefrontal cortex (DLPFC) and the cathode will be placed over the right supraorbital cortex. This is the standard 1 anode by 1 cathodal convention. Stimulation will last 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- High Definition (HD)-tDCS stimulation (Experimental): Transcranial Direct Current Stimulation:
  The anode will be placed over the left DLPFC and 4 cathodes will be placed surrounding the anode. This is the 4 cathode by 1 anode HD-tDCS montage for more focal stimulation. Stimulation will last 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS sham stimulation (Sham Comparator): Transcranial Direct Current Stimulation:
  The anode will be placed over the left DLPFC and the cathode over the right supraorbital cortex. A short stimulation will be given to the subjects that will mimic the sensation of an actual stimulation but will last much shorter. The session will still last 20 minutes in total to blind both subjects and investigators.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — TDCS involves sending a weak electrical current to the brain to modulate brain functions.
  Other Names: Neuroelectrics Starstim

SUMMARY:
The purpose of this study is to test the effects of tDCS (Transcranial Direct Current Stimulation) on stroke patients with working memory problems.

DETAILED DESCRIPTION:
After having a stroke, people often have trouble remembering to do something, solving problems, or following conversations. They can also have trouble concentrating, following instructions, and multitasking. These can all due to the stroke affecting a brain function called "working memory". Working memory is defined as the ability to hold a thought in one's mind for a few seconds in order to remember a task or solve a problem. People have difficulty returning to their normal lives because of these working memory problems. Currently, there no proven medical treatments for working memory problems.

Transcranial direct current stimulation (tDCS) is a painless, noninvasive brain stimulation technique that has been shown in some studies to improve working memory in healthy subjects. TDCS involves sending a weak electrical current through the head, thereby exciting the brain underneath. TDCS is not an FDA-approved treatment for any condition, but previous trials have shown it may benefit movement and language recovery after stroke, as well as improve thinking ability. Studies have shown tDCS to be very safe with no serious adverse events in over 10,000 subjects studied.

This pilot study will involve four visits to Stony Brook University Hospital. The first is a baseline session where subjects perform all outcome measures but no tDCS is performed other than for familiarization. The other three sessions are the stimulation sessions where subjects undergo the intervention for 20 minutes to test tDCS effects on the outcome measures. The effects of tDCS for a single session are expected to only last for few hours. Subjects will be receiving all three different types of stimulation. If this study finds a short term benefit of tDCS for post-stroke working memory deficits, it will support a full clinical trial where multiple sessions of tDCS will be given and may provide a long-term benefit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke and radiographically proven ischemic or hemorrhagic stroke (MRI required for ischemic stroke, CT sufficient for hemorrhagic stroke).
* Subject reports a decline in attention or short-term memory that began at the time of their stroke.
* Stroke occurred at least one month prior to first stimulation session.
* Ability to provide informed consent.
* Speak English (required for performing the cognitive tests)

Exclusion Criteria:

* Any other brain disease that can affect cognition (e.g., multiple sclerosis, dementia).
* Active mental illness such as depression or anxiety
* Large stroke involving cortex under the stimulation site (using subject provided CT or MRI).
* Currently taking any drugs that are sodium and/or calcium channel blockers not including amlodipine. This includes some seizure medications along with nicardipine, nifedipine, nimodipine, verapamil and diltiazem.
* Any history of epilepsy.
* Subject report of recent drug or alcohol abuse - within the past year.
* Subject report of pregnant or breastfeeding.
* Moderate to severe aphasia preventing subject from communicating fully.
* Any pacemakers, intracranial electrodes, implanted defibrillators, or any other electrical implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in Cognitive Test Battery | before and after each stimulation within 2 hours.
  A series of cognitive tests will be conducted before and after each stimulation. The tests will include a n-back test (0,1,2), a delayed recognition task, and a number capacity task.

SECONDARY OUTCOMES:
Changes in Auditory Digit Span Test | at baseline, once immediately after stimulation, one time in the evening of the session day and then one more time the day after the session
  An auditory digit span test (forward and backward) will be asked over phone 4 times.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Goldfine, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845